CLINICAL TRIAL: NCT03613870
Title: A Prospective, Randomized, Parallel Study to Evaluate the Effectiveness of PermeaDerm® and Mepilex-Ag® in Promoting Healing of Partial-thickness Burn Wounds
Brief Title: PermeaDerm® vs. Mepilex-Ag® in Promoting Healing of Partial-thickness Burn Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively closed prior enrollment of participants.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0315
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Partial-thickness Burn
Keywords: PermeaDerm, Mepilex Ag, partial thickness burn wounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PermeaDerm (Active Comparator): Participants receive PermeaDerm dressing for wound treatment until wounds have healed completely
  Interventions: Device: PermeaDerm
- Mepilex Ag (Active Comparator): Participants receive Mepilex Ag dressing for wound treatment until wounds have healed completely
  Interventions: Device: Mepilex Ag

INTERVENTIONS:
Device: PermeaDerm — Wound treatment with PermeaDerm
  Arms: PermeaDerm
Device: Mepilex Ag — Wound treatment with Mepilex Ag
  Arms: Mepilex Ag

SUMMARY:
The purpose of this study is to compare the effectiveness of the wound dressings currently used at our institution for partial-thickness burn wounds: PermeaDerm® (PermeaDerm, Inc., Carlsbad, California, USA) and silver impregnated foam dressing (Mepilex Ag®, Health Care, Göteborg, Sweden)

DETAILED DESCRIPTION:
In this prospective, randomized parallel study, the effectiveness of the wound dressings currently used at our institution for partial-thickness burn wounds will be compared: PermeaDerm®, and silver coated foam dressing Mepilex Ag®.This study is therefore considered a minimal risk study. Procedures related to research apart from randomization to one of the dressings, will include review of medical records, non-invasive wound and scar assessments and additional photographs.

60 patients with partial thickness burns meeting the inclusion criteria of the study will be enrolled to receive either PermeaDerm® (n=30) or silver coated foam dressing (Mepilex Ag®; n=30) in an outpatient or observational setting.

Prior to placement of wound dressings, baseline assessments of wound size and burn depth will be performed by the experienced physician and documented using photography and when indicated laser Doppler (Moor Laser Speckle®, Moor Instruments, Devon, UK) measurements. Time to heal will be defined as the time after which complete re-epithelialization is reached and PermeaDerm® detaches or there are no more changes of Mepilex Ag® needed. Secondary goals of the study are to assess pain, and scarring associated with the use of the different dressings in our burn patients, as well as to assess cost-effectiveness of the therapy.

Pain will be assessed at every patient visit using visual analog scale (VAS) or Wong-Baker FACES respectively; mid and long-term scar development is assessed at approximately 1 and 6 months after enrollment in the study using Patient and Observer Scar Assessment Scale (POSAS) and DermaLab Combo® (Cortex Technology, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Superficial partial thickness burn injury due to flame burn, scald injury or contact burn that does not require excision and grafting
* Total Body Surface Area burned (TBSA) total ≤30 %
* Admission within 72 hours of burn injury
* Non-infected wound as diagnosed by the attending physician upon admission
* Treated as an outpatient or in an observational setting

Exclusion Criteria:

* Patient younger than 6 months
* Causes other than contact burn, flame or scald injuries (i.e., electrical, chemical or frostbite)
* Admission time greater than 72 hours after the injury
* Wounds noted to be infected at admission
* Previous treatment efforts such as previous debridement, silver sulfadiazine ointment or other pseudo eschar-forming topical agents
* Pregnancy/lactation

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Time to heal | up to 3 weeks after injury
  Time until wound is complete healed in days. A wound is considered as completely healed, when either PermeaDerm detaches on its own or no more dressings need to be applied in the Mepilex group. This time point is defined when approximately 95% of the wound shows epithelialization as determined by an experienced burn surgeon.

SECONDARY OUTCOMES:
Pain assessment using Visual Analog Pain Scale (VAS) or Wong-Baker FACES pain rating scales (age dependent) | Changes over first 30 days post injury, using regression modeling for analysis.
  Pain assessment using Visual Analog Scale rating Pain scores ranging from 0-10 (8 years and older) OR Wong-Baker FACES Pain Rating Scale (3-7 years old). FACES stands for faces, since this rating scale shows faces from very happy to very unhappy. It ranges also from 0-10. Higher values indicating greater pain. The 0-10 scores for each scale are equivalent.
Scar assessment with Patient and Observer Assessment Scale (POSAS) | at 1 month post injury
  Using Patient and Observer Scar Assessment Scale POSAS, what is a composite score that is rating the overall appearance of the scar, based on each single score for rating vascularity, pigmentation, thickness, relief, pliability, surface. Every subscore ranges from 1-10. The composite score is calculated as an average of the subscores. Higher numbers mean worse scarring.
Scar assessment with Patient and Observer Assessment Scale (POSAS) | at 6 months post injury
  Using Patient and Observer Scar Assessment Scale POSAS, what is a composite score that is rating the overall appearance of the scar, based on each single score for rating vascularity, pigmentation, thickness, relief, pliability, surface. Every subscore ranges from 1-10. The composite score is calculated as an average of the subscores. Higher numbers mean worse scarring.
Scarring with DermaLab Combo device: Viscoelasticity | at 1 month post injury
  Measured through negative suction and retraction time.
Scarring with DermaLab Combo device: Viscoelasticity | at 6 months post injury
  Measured through negative suction and retraction time.
Scarring with DermaLab Combo device: Hydration | at 1 month post injury
  Measured based on skin conductance.
Scarring with DermaLab Combo device: Hydration | at 6 months post injury
  Measured based on skin conductance.
Scarring with DermaLab Combo device: Pigmentation | at 1 month post injury
  Measured based on light absorption of melanin and erythema
Scarring with DermaLab Combo device: Pigmentation | at 6 months post injury
  Measured based on light absorption of melanin and erythema
Scarring with DermaLab Combo device: Trans epithermal water loss | at 1 month post injury
  Measuring evaporation in g/meter square/hour
Scarring with DermaLab Combo device: Trans epithermal water loss | at 6 months post injury
  Measuring evaporation in g/meter square/hour
Rate of Infection | at 1 month post burn
  Defined as bacterial growth of >10 to power of 5 in swab. Only taken when infection suspected.
Cost-effectiveness | at 1 month post burn
  Number of dressing changes required until healing versus respective product costs (costs per cm square)

CONTACTS AND LOCATIONS:
Overall Officials: Ludwik K Branski, MD, Principal Investigator — The University of Texas Medical Branch, Galveston

IPD SHARING:
Plan to Share IPD: No
data won't be shared